CLINICAL TRIAL: NCT04905537
Title: Study on Early Genetic Screening and Precise Strategy of Neonatal Critical Illness
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: International Peace Maternity and Child Health Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Children's Medical Center (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU15
Record Dates: First submitted 2021-05-25; First posted 2021-05-27 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Genetic Screening; Hereditary Disease; Newborn; Stillbirth
MeSH Terms: conditions — Genetic Diseases, Inborn; Stillbirth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The researchers retained the neonates', infants' or stillbirths' 2ml peripheral blood, cord blood, amniotic fluid, muscle or saliva as a biological sample for gene screening.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sick Neonates or Stillbirth: Infants and their parents enrolled through Neonatal Intensive Care Unit or stillbirths through Obstetrics Department of member hospitals who are un-randomized to receive genomic sequencing. Results disclosure sessions will include a discussion of: family history report, results from standard newborn screening, any potentially medically relevant findings from the baby's medical history/ physical exam, and the results of the genomic sequencing report.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — It's only observational study. No interventions.

SUMMARY:
The researchers hope to establish an overall program of early genetic screening for neonatal critical illness in China, and to develop precise intervention strategies to assist clinical diagnosis and treatment of hereditary critical illness.

DETAILED DESCRIPTION:
Reducing the rate of neonatal death and disability is an important part of health education in China, and genetic diseases are an important cause of neonatal death. At present, with the development of life support platform technology, the treatment level of critically ill newborns has been rapidly improved. How to quickly diagnose and early precise intervention is the key to further break through the diagnosis and treatment of genetic diseases. Based on the "neonatal genome project" carried out in the early stage, the research group based on the genetic diagnosis results of over 10000 cases of neonatal critical illness cohort, studied the genetic disease spectrum of neonatal critical illness in line with the actual situation in China. In terms of detection technology, based on the second-generation sequencing technology, we established a critical illness screening gene sequencing combination including 300 genes; In the aspect of data analysis, an intelligent analysis process integrating clinical phenotype and gene sequencing data was established; In terms of clinical diagnosis and treatment, we cooperated with 5 maternity and children's hospitals in Shanghai to carry out multi center clinical verification, and formed the implementation plan of early universal genetic screening for neonatal critical illness. Through this project, we will carry out genetic disease screening research on neonatal critical diseases, focus on typical clinical manifestations such as encephalopathy, immunodeficiency, metabolic diseases, and carry out molecular autopsy on neonatal death cases to identify potential genetic causes, so as to provide basis for the research of corresponding early precise intervention strategies, and achieve the purpose of reducing neonatal death and disability rate.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age less than 100 days;
* Perinatal death after 20 weeks of gestation (more than 500 g)
* Can be retained biological samples for genetic screening;
* Biological parent or guardian's informed consent.

Exclusion Criteria:

* Reluctance of parents to use genetic sequencing data for subsequent research;
* Parents under 18 years of age or incapacitated for decision-making;
* subjects older than 100 days;
* Perinatal death less than 20 weeks of gestation or weight less than 500 g;
* Inherited metabolic diseases with chromosomal abnormalities;
* Multiple pregnancies;
* Lack of access to biological samples from which DNA can be extracted;
* Failure to sign informed consent.

Max Age: 100 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects were all from all the member organizations participating in this research. They were hospitalized in the neonatal department or stillbirth in obstetrics department of each member hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gene Mutation | In 3 months after receipt of the samples
  To detect the mutation and characterize the genetic architecture and risk variants (911 variants of 146 genes, for example, AGT, AGTR1, CA12, CD2AP et al) of subjects using different genomic methods

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Yang L, Liu X, Li Z, Zhang P, Wu B, Wang H, Hu L, Cheng G, Wang L, Zhou W. Genetic aetiology of early infant deaths in a neonatal intensive care unit. J Med Genet. 2020 Mar;57(3):169-177. doi: 10.1136/jmedgenet-2019-106221. Epub 2019 Sep 9. PMID 31501239
- [Background] Stevenson DA, Carey JC. Contribution of malformations and genetic disorders to mortality in a children's hospital. Am J Med Genet A. 2004 May 1;126A(4):393-7. doi: 10.1002/ajmg.a.20409. PMID 15098237
- [Background] Willig LK, Petrikin JE, Smith LD, Saunders CJ, Thiffault I, Miller NA, Soden SE, Cakici JA, Herd SM, Twist G, Noll A, Creed M, Alba PM, Carpenter SL, Clements MA, Fischer RT, Hays JA, Kilbride H, McDonough RJ, Rosterman JL, Tsai SL, Zellmer L, Farrow EG, Kingsmore SF. Whole-genome sequencing for identification of Mendelian disorders in critically ill infants: a retrospective analysis of diagnostic and clinical findings. Lancet Respir Med. 2015 May;3(5):377-87. doi: 10.1016/S2213-2600(15)00139-3. Epub 2015 Apr 27. PMID 25937001
- [Background] Daoud H, Luco SM, Li R, Bareke E, Beaulieu C, Jarinova O, Carson N, Nikkel SM, Graham GE, Richer J, Armour C, Bulman DE, Chakraborty P, Geraghty M, Lines MA, Lacaze-Masmonteil T, Majewski J, Boycott KM, Dyment DA. Next-generation sequencing for diagnosis of rare diseases in the neonatal intensive care unit. CMAJ. 2016 Aug 9;188(11):E254-E260. doi: 10.1503/cmaj.150823. Epub 2016 May 30. PMID 27241786
- [Background] Amberger JS, Hamosh A. Searching Online Mendelian Inheritance in Man (OMIM): A Knowledgebase of Human Genes and Genetic Phenotypes. Curr Protoc Bioinformatics. 2017 Jun 27;58:1.2.1-1.2.12. doi: 10.1002/cpbi.27. PMID 28654725
- [Background] Ceyhan-Birsoy O, Murry JB, Machini K, Lebo MS, Yu TW, Fayer S, Genetti CA, Schwartz TS, Agrawal PB, Parad RB, Holm IA, McGuire AL, Green RC, Rehm HL, Beggs AH; BabySeq Project Team. Interpretation of Genomic Sequencing Results in Healthy and Ill Newborns: Results from the BabySeq Project. Am J Hum Genet. 2019 Jan 3;104(1):76-93. doi: 10.1016/j.ajhg.2018.11.016. PMID 30609409
- [Background] Berg JS, Agrawal PB, Bailey DB Jr, Beggs AH, Brenner SE, Brower AM, Cakici JA, Ceyhan-Birsoy O, Chan K, Chen F, Currier RJ, Dukhovny D, Green RC, Harris-Wai J, Holm IA, Iglesias B, Joseph G, Kingsmore SF, Koenig BA, Kwok PY, Lantos J, Leeder SJ, Lewis MA, McGuire AL, Milko LV, Mooney SD, Parad RB, Pereira S, Petrikin J, Powell BC, Powell CM, Puck JM, Rehm HL, Risch N, Roche M, Shieh JT, Veeraraghavan N, Watson MS, Willig L, Yu TW, Urv T, Wise AL. Newborn Sequencing in Genomic Medicine and Public Health. Pediatrics. 2017 Feb;139(2):e20162252. doi: 10.1542/peds.2016-2252. Epub 2017 Jan 17. PMID 28096516
- [Background] Sanford EF, Clark MM, Farnaes L, Williams MR, Perry JC, Ingulli EG, Sweeney NM, Doshi A, Gold JJ, Briggs B, Bainbridge MN, Feddock M, Watkins K, Chowdhury S, Nahas SA, Dimmock DP, Kingsmore SF, Coufal NG; RCIGM Investigators. Rapid Whole Genome Sequencing Has Clinical Utility in Children in the PICU. Pediatr Crit Care Med. 2019 Nov;20(11):1007-1020. doi: 10.1097/PCC.0000000000002056. PMID 31246743